CLINICAL TRIAL: NCT04088929
Title: A Dose Controlled Diabetic Neuropathic Pain Study Using Non-Intoxicating Cannabidiol in a Rapidly Dissolvable Sublingual Tablet
Brief Title: The Use of a Water Soluble Under the Tongue (Sublingual) CBD Tablet for Treating Pain Associated With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pure Green (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-19-002
Record Dates: First submitted 2019-09-10; First posted 2019-09-13 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Neuropathies
Keywords: Pain; Neuropathy; Neuropathic Pain; Diabetes
MeSH Terms: conditions — Diabetic Neuropathies; Pain; Neuralgia; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBD for Treatment of Diabetic Neuropathic Pain (Experimental): Patients are instructed to take 3 total tablets a day, under the tongue, six hours apart for three weeks. Patients are to enter their pain scale score into the smartphone app as instructed during the initial site visit. Patients are to enter into the notes section of the app any additional information such as side effects (positive or negative), medication changes.
  Interventions: Drug: CBD

INTERVENTIONS:
Drug: CBD — A water-soluble sublingual tablet containing 20 mg of cannabidiol (CBD) and 0.1 mg of a proprietary blend of terpenes.

SUMMARY:
Use of Cannabidiol for the treatment of Diabetic Neuropathic Pain.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 21 years of age;
2. Subject has a diagnosis of chronic diabetic neuropathic pain condition as determined by the subject's health care or allied health provider for which medications other than cannabis, cannabinoids, or cannabis-based medicines are currently utilized;
3. Subject has a 7-day average pain scale score (recorded during the screening period) of ≥ 5;
4. If female, subject is postmenopausal (> 1 year), surgically sterile, or practicing an approved method of birth control throughout the study and for 5 months (150 days) after the last dose of study drug;
5. If female and of childbearing potential, subject has a denied pregnancy and has no desire to become pregnant throughout the duration of the study;
6. Subject is willing and able to provide his/her written informed consent to participate in the study as stated in the informed consent document;
7. Subject has access to a smart phone and knows how to use smart phone applications.

Exclusion Criteria:

1. Subject is pregnant or lactating;
2. Subject has an allergy to cannabis, the Cannabaceae plant family (e.g., hemp, hops, hackberry), PEA, terpenes, peppermint;
3. Subject has a known allergy to active or inert ingredients of Pure Green tablets;
4. Subject is currently treating their pain with cannabis, cannabinoids, cannabis-base medicine;
5. Subject is taking a concomitant medication or treatment that would complicate use or interpretation of the study drug's effects (examples include: Cannabis or any cannabinoid products; Any drug or herbal product that influences the endocannabinoid system (ECS));
6. Subject is taking marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD for at least 30 days prior to this study., and does not promise to not take marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD while participating in this study;
7. Subject is currently being treated with antibiotics for sinus, throat, or lung infections;
8. Subject has shortness of breath associated with allergies;
9. Subject has uncontrolled asthma;
10. Subject has a fever and/or productive cough;
11. Subject does not have access to a smart phone or does not know how to use a smart phone application.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Impact of Pure Green CBD tablets on diabetic neuropathy pain using a daily self-reported pain scale score. | Three Weeks
  To evaluate the safety and efficacy of Pure Green CBD sublingual tablets for the treatment of chronic diabetic neuropathic pain patients by evaluating their daily pain scale score reported as 0-10 where 0 is no pain and 10 is the worst pain possible as self-reported with every dose taken by the patient in the smart phone app. The objective is to reduce the patients average daily pain scale score to less than 5.

SECONDARY OUTCOMES:
Impact of Pure Green CBD tablets on the quality of life of Diabetic Neuropathy Patients | Three Weeks
  To evaluate the impact of Pure Green CBD sublingual tablets on the quality of life of diabetic neuropathy patients measured by World Health Organization's quality of life questionnaire, . The objective is to examine quality of life metrics: overall quality of life and general health, physical health, psychological, social, and environment as measured on a 1-5 scale before and after the study.
Impact of Pure Green CBD tablets on sleep improvement of Diabetic Neuropathy Patients | Three weeks
  The Pittsburgh Sleep Quality Index will be used to compare pre and post Pure Green CBD tablet study on sleep changes. Patients will be asked questions before beginning the study and after completion.
Impact of Pure Green CBD tablets on anxiety of Diabetic Neuropathy Patients | Three Weeks
  The Hamilton Anxiety rating scale questionnaire will be administered before the study begins and after completion to examine the impact of Pure Green CBD tablets on anxiety in diabetic neuropathy pain patients. The scale of 0-4 will be used where 0 is no anxiety present and 4 is very severe anxiety.
Impact on the use of sublingual tablets as the route of administration | Three Weeks
  To explore the impact of sublingual administration on patient compliance by evaluating the number of tablets taken per day as entered by the patients into the smart phone app.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kimless, M.D., Principal Investigator — Pure Green, LLC
Locations (1):
- Dr. Nakadar's Office, Sterling Heights, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quattrini C, Tesfaye S. Understanding the impact of painful diabetic neuropathy. Diabetes Metab Res Rev. 2003 Jan-Feb;19 Suppl 1:S2-8. doi: 10.1002/dmrr.360. PMID 12577252
- [Background] Callaghan BC, Cheng HT, Stables CL, Smith AL, Feldman EL. Diabetic neuropathy: clinical manifestations and current treatments. Lancet Neurol. 2012 Jun;11(6):521-34. doi: 10.1016/S1474-4422(12)70065-0. Epub 2012 May 16. PMID 22608666
- [Background] Argoff CE, Cole BE, Fishbain DA, Irving GA. Diabetic peripheral neuropathic pain: clinical and quality-of-life issues. Mayo Clin Proc. 2006 Apr;81(4 Suppl):S3-11. doi: 10.1016/s0025-6196(11)61474-2. PMID 16608048
- [Background] Sadosky A, Mardekian J, Parsons B, Hopps M, Bienen EJ, Markman J. Healthcare utilization and costs in diabetes relative to the clinical spectrum of painful diabetic peripheral neuropathy. J Diabetes Complications. 2015 Mar;29(2):212-7. doi: 10.1016/j.jdiacomp.2014.10.013. Epub 2014 Nov 8. PMID 25498300
- [Background] Gordois A, Scuffham P, Shearer A, Oglesby A, Tobian JA. The health care costs of diabetic peripheral neuropathy in the US. Diabetes Care. 2003 Jun;26(6):1790-5. doi: 10.2337/diacare.26.6.1790. PMID 12766111
- [Background] Singh R, Kishore L, Kaur N. Diabetic peripheral neuropathy: current perspective and future directions. Pharmacol Res. 2014 Feb;80:21-35. doi: 10.1016/j.phrs.2013.12.005. Epub 2013 Dec 25. PMID 24373831
- [Background] Boulton AJ: Management of Diabetic Peripheral Neuropathy. Clinical Diabetes. 2005;23(1):9-15.
- [Background] Wallace MS, Marcotte TD, Umlauf A, Gouaux B, Atkinson JH. Efficacy of Inhaled Cannabis on Painful Diabetic Neuropathy. J Pain. 2015 Jul;16(7):616-27. doi: 10.1016/j.jpain.2015.03.008. Epub 2015 Apr 3. PMID 25843054
- [Background] Bridges D, Ahmad K, Rice AS. The synthetic cannabinoid WIN55,212-2 attenuates hyperalgesia and allodynia in a rat model of neuropathic pain. Br J Pharmacol. 2001 Jun;133(4):586-94. doi: 10.1038/sj.bjp.0704110. PMID 11399676
- [Background] De Vry J, Denzer D, Reissmueller E, Eijckenboom M, Heil M, Meier H, Mauler F. 3-[2-cyano-3-(trifluoromethyl)phenoxy]phenyl-4,4,4-trifluoro-1-butanesulfonate (BAY 59-3074): a novel cannabinoid Cb1/Cb2 receptor partial agonist with antihyperalgesic and antiallodynic effects. J Pharmacol Exp Ther. 2004 Aug;310(2):620-32. doi: 10.1124/jpet.103.062836. Epub 2004 May 12. PMID 15140913
- [Background] Abrams DI, Jay CA, Shade SB, Vizoso H, Reda H, Press S, Kelly ME, Rowbotham MC, Petersen KL. Cannabis in painful HIV-associated sensory neuropathy: a randomized placebo-controlled trial. Neurology. 2007 Feb 13;68(7):515-21. doi: 10.1212/01.wnl.0000253187.66183.9c. PMID 17296917
- [Background] Ware MA, Wang T, Shapiro S, Robinson A, Ducruet T, Huynh T, Gamsa A, Bennett GJ, Collet JP. Smoked cannabis for chronic neuropathic pain: a randomized controlled trial. CMAJ. 2010 Oct 5;182(14):E694-701. doi: 10.1503/cmaj.091414. Epub 2010 Aug 30. PMID 20805210
- [Background] Wilsey B, Marcotte T, Deutsch R, Gouaux B, Sakai S, Donaghe H. Low-dose vaporized cannabis significantly improves neuropathic pain. J Pain. 2013 Feb;14(2):136-48. doi: 10.1016/j.jpain.2012.10.009. Epub 2012 Dec 11. PMID 23237736
- [Background] Wilsey B, Marcotte T, Tsodikov A, Millman J, Bentley H, Gouaux B, Fishman S. A randomized, placebo-controlled, crossover trial of cannabis cigarettes in neuropathic pain. J Pain. 2008 Jun;9(6):506-21. doi: 10.1016/j.jpain.2007.12.010. Epub 2008 Apr 10. PMID 18403272
- [Background] Johnson JR, Burnell-Nugent M, Lossignol D, Ganae-Motan ED, Potts R, Fallon MT. Multicenter, double-blind, randomized, placebo-controlled, parallel-group study of the efficacy, safety, and tolerability of THC:CBD extract and THC extract in patients with intractable cancer-related pain. J Pain Symptom Manage. 2010 Feb;39(2):167-79. doi: 10.1016/j.jpainsymman.2009.06.008. Epub 2009 Nov 5. PMID 19896326
- [Background] De Gregorio D, McLaughlin RJ, Posa L, Ochoa-Sanchez R, Enns J, Lopez-Canul M, Aboud M, Maione S, Comai S, Gobbi G. Cannabidiol modulates serotonergic transmission and reverses both allodynia and anxiety-like behavior in a model of neuropathic pain. Pain. 2019 Jan;160(1):136-150. doi: 10.1097/j.pain.0000000000001386. PMID 30157131